CLINICAL TRIAL: NCT04930601
Title: HBP Synchrony Using ECG Belt
Brief Title: HIS Bundle Pacing Synchrony Comparing HIS Pacing to Intrinsic Conduction While Using the Medtronic ECG Belt System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SAMBIT MONDAL (Other)
Responsible Party: Sponsor-Investigator, SAMBIT MONDAL, MD, Orlando Cardiac and Vascular Specialists
Organization: Orlando Cardiac and Vascular Specialists (Other)
Other Study IDs: OSCMondal062021
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: HBP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
The HBP Synchrony Using ECG Belt study is a prospective, non-randomized single site physician-initiated research study. The study will collect ECG Belt data from up to 30 subjects at one single center. The target population will include subjects with a currently implanted Medtronic cardiac implantable device who have a HIS placed lead. The purpose of the study is to characterize the electrical dispersion using the ECG Belt provided by Medtronic in patients who have a HIS placed lead and understanding the amount of synchrony with intrinsic conduction compared to HIS pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patient has previously been implanted with a Medtronic IPG/ICD and a HIS placed RV lead
* Patient has intrinsic AV conduction
* Normal EF, defined as EF >50%, as shown on recent echo within last 12 months
* Patient is willing and able to comply with the protocol
* Patient is 18 years of age or older

Exclusion Criteria:

●Patient is ventricular pacer dependent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population will include subjects with normal EF who have a Medtronic device and a HIS placed RV lead. In addition, we will include subjects who have intact AV conduction.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the electrical dispersion using SDAT | 1 year
  Characterize the electrical dispersion between intrinsic to both Selective HIS pacing and Non-Selective HIS pacing using Standard Deviation Activation Timing of the ECG Belt system.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Cardiac & Vascular Specialists, Altamonte Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided